CLINICAL TRIAL: NCT05454332
Title: The Caffeine Therapy in the Fetal to Neonatal Transition in Preterms
Brief Title: The Caffeine Therapy in the Fetal to Neonatal Transition
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Gabriela Scholer Trindade, Doctor, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021-0463
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-05

CONDITIONS: Mechanical Ventilation Complication; Caffeine; Ventilator Lung; Newborn
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Caffeine Group (Experimental): Group administering caffeine in the first 2 hours of life. Patients in the early caffeine group will receive an attack dose of caffeine 20 mg/kg and begin maintenance dose 10 mg/kg/day.
  Interventions: Drug: Early Caffeine administration
- Control Group (Active Comparator): Patients in the late caffeine group, receive bolus of saline solution in the first 2 hours of life, starting, at 24 hours of life, the caffeine-loading dose 20 mg/kg and after maintenance dose 10mg/kg/day.
  Interventions: Other: Control Group

INTERVENTIONS:
Drug: Early Caffeine administration — Blinding will be done with the administration of saline solution. Patients in the early caffeine group will receive an attack dose of caffeine 20 mg/kg and begin maintenance dose 10 mg/kg/day. Patients in the late caffeine group, receive bolus of saline solution in the first 2 hours of life, starting, at 24 hours of life, the caffeine-loading dose 20 mg/kg and after maintenance dose 10mg/kg/day. The medical team will prescribe the medication, and the pharmacy will be responsible for randomly dispensing the caffeine or saline solution. The pharmacy will prepare syringes with the medication or saline solution identified by a code referring to the randomization without identifying which solution is being administered. The syringes will be sent to the neonatal ICU and will be administered according to the physician's prescription. The administration will be blinded.
  Arms: Early Caffeine Group
Other: Control Group — Blinding will be done with the administration of saline solution. Patients in the early caffeine group will receive an attack dose of caffeine 20 mg/kg and begin maintenance dose 10 mg/kg/day. Patients in the late caffeine group, receive bolus of saline solution in the first 2 hours of life, starting, at 24 hours of life, the caffeine-loading dose 20 mg/kg and after maintenance dose 10mg/kg/day. The medical team will prescribe the medication, and the pharmacy will be responsible for randomly dispensing the caffeine or saline solution. The pharmacy will prepare syringes with the medication or saline solution identified by a code referring to the randomization without identifying which solution is being administered. The syringes will be sent to the neonatal ICU and will be administered according to the physician's prescription. The administration will be blinded.
  Arms: Control Group

SUMMARY:
Introduction: The caffeine is used in the treatment for apnea of prematurity and it has several positive effects in the neurodevelopment of preterm babies. There are innumerable observational studies suggesting that initiating caffeine in the first hours of life may offer more benefits in the reduction of the necessity of intubation and in ventilation time. It is necessary to expand further research on the best time to start caffeine, which may improve the quality of care for premature infants.

Objective: To evaluate the benefits of caffeine administration in the first two hours of life compared to administration at 24 hours of life in premature patients on noninvasive mechanical ventilation with birth weights less than 1250 grams.

Methodology: Preterm newborn patients with birth weight < 1250 grams born at Hospital de Clínicas de Porto Alegre who are not intubated in the delivery room will be included. Patients will be randomized into two groups. One arm of the study will receive caffeine at 2 hours of age and the other arm will receive caffeine at 24 hours of age (control). Patients in the control group will receive 0.9% SF at 2 hours of life in order to keep the study blinded. The following outcomes will be evaluated: need for intubation, time on invasive and non-invasive mechanical ventilation, BPD, necrotizing enterocolitis, need for ROP treatment, PDA with hemodynamic repercussions, peri-intraventricular hemorrhage, leukomalacia and death. The sample size calculation is 50 patients, 25 in each arm.

Expected Results: It is expected to find a 43% reduction in the need for intubation in preterm infants who receive caffeine in the first two hours of life compared to administration at 24 hours of life. It is also expected to find a reduction in mechanical ventilation time, in addition to a possible reduction in negative outcomes associated with prematurity.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborns with birth weight less than 1250 grams
* Who are not intubated in the delivery room

Exclusion Criteria:

* Premature newborns from other hospitals
* Presence of a major congenital malformation or genetic syndrome

Max Age: 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Necessity of intubation | first week of life
  Noninvasive ventilation failure will be defined as intubation in the first seven days of life with the need for invasive ventilation for at least 24 hours.

SECONDARY OUTCOMES:
mechanical ventilation time | until first successful extubation (followed up at least until 36 weeks of corrected age, discharge or death)
  Mechanical ventilation time will be counted until first successful extubation (at least 24 hours extubated)
Number of Participants with Bronchopulmonary dysplasia | followed up at least until 36 weeks of corrected age, discharge or death.
  Bronchopulmonary dysplasia will be defined as need for O2 or ventilatory support at 36 weeks corrected gestational age.
Number of Participants with Intracranial hemorrhage | followed up at least until 36 weeks of corrected age, discharge or death.
  Intracranial hemorrhage will be defined as intracranial hemorrhage grade 3.
Number of Participants with Retinopathy of prematurity | followed up at least until 36 weeks of corrected age, discharge or death.
  Retinopathy of prematurity will be defined with ROP requiring treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil